CLINICAL TRIAL: NCT02613585
Title: Tick-borne Illness and Clothing Study of Rhode Island
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of Rhode Island (Other); East Carolina University (Other); National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 15-1770; R01OH010791 (NIH)
Record Dates: First submitted 2015-11-20; First posted 2015-11-24 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-02

CONDITIONS: Tick Bites; Tick-borne Diseases
MeSH Terms: conditions — Tick Bites; Tick-Borne Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Permethrin Impregnated Clothing (Experimental): Uniforms and work clothing (including pants, shorts, shirts, socks, and hats) treated with long-lasting permethrin by Insect Shield.
  Interventions: Other: Permethrin Impregnated Clothing
- Untreated Clothing (No Intervention): Uniforms and work clothing sent to Insect Shield, washed and refolded (no permethrin applied).

INTERVENTIONS:
Other: Permethrin Impregnated Clothing — Uniforms and work clothing treated with permethrin according to proprietary process used by Insect Shield, Inc.
  Other Names: Insect Shield
  Arms: Permethrin Impregnated Clothing

SUMMARY:
Lyme and other tick-borne diseases pose a significant health threat to outdoor workers. This study is a double-blind randomized controlled trial of outdoor workers in Rhode Island and the surrounding area that will address the following study aims: 1) Evaluate the effectiveness of LLPI clothing in preventing tick bites among outdoor workers in Lyme endemic areas; 2) Measure the urine levels of permethrin metabolites in study subjects; and 3) Measure the loss over time of knockdown activity against ticks and of permethrin in LLPI clothing.

DETAILED DESCRIPTION:
Lyme and other tick-borne diseases pose a significant health threat to outdoor workers. In a double-blind randomized controlled trial (RCT) in North Carolina outdoor workers, the investigators previously showed that long-lasting permethrin-impregnated (LLPI) clothing provided >80% protection for one year against Lone Star tick bites among outdoor workers in North Carolina. But there are three issues that need to be addressed before this finding can be translated into policy: 1) Do LLPI clothing protect against black legged ticks, the vector for Lyme disease, babesiosis and anaplasmosis? 2) What levels of permethrin and its metabolites are absorbed, and are they potentially toxic? 3) Why did the LLPI clothing in our previous study lose efficacy after a year?

Participants: The investigators will recruit 250 outdoor workers. The investigators anticipate recruiting 80, 80, 40,30, and 20 participants from NationalGrid, the RI Department of Environmental Management, the Massachusetts Department of Conservation & Recreation, the National Park Service, and the US Fish & Wildlife Service.

Procedures (methods): This will be a randomized controlled trial. All study subjects will fill out weekly tick logs, collect attached ticks for later speciation and pathogen detection, and submit annual serum samples to test for exposure to tick-borne pathogens. A randomly selected subset of 60 subjects also will be asked to submit urine samples for permethrin metabolite analysis at several time points during follow-up. An additional randomly selected subset (n=30) will be asked to submit worn items of clothing for tick knockdown testing and permethrin content analysis at the end of the first and second years of field testing.

The results of this study could help protect hundreds of thousands of outdoor workers with exposure to ticks and tick-borne pathogens.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age,
* spending an average of 10 or more hours of outdoor work per week during peak tick season, and
* completion of written informed consent.

Exclusion Criteria:

* pregnancy or a planned pregnancy during the follow-up period (since exposure to an insecticide is involved),
* non-English speakers, or
* having a known allergy or sensitivity to insecticides

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Number of Work Related Tick Bites Per Week | Weekly for two years
  Reported tick bites, defined as ticks attached to or embedded in the skin.

SECONDARY OUTCOMES:
Change in permethrin metabolite levels after 3 weeks | Enrollment to 3 weeks after study initiation
  Permethrin metabolites measured in urine, compared to baseline prior to wearing clothing.
Change in permethrin metabolite levels after 1 year | Enrollment to end of study year 1
  Metabolites measured in urine, compared to baseline prior to wearing clothing.
Change in concentration of permethrin in clothing after 1 year | Enrollment to end of study year 1
  Measurement of the chemical concentration of clothing samples after study year 1, compared against concentration of a newly treated clothing sample.
Change in concentration of permethrin in clothing after 2 years | Enrollment to 2 years after study initiation
  Measurement of the chemical concentration of clothing samples after study year 2, compared against concentration of a newly treated clothing sample.
Change in tick repellency after 1 year | Enrollment to 1 year after study initiation
  Measurement of the tick repellency ("knockdown activity") of clothing samples after study year 1, compared against concentration of a newly treated piece of clothing sample.
Change in tick repellency after 2 years | Enrollment to 2 years after study initiation
  Measurement of the tick repellency ("knockdown activity") of clothing samples after study year 2, compared against concentration of a newly treated piece of clothing sample.
Pathogen seroconversion in study year 1 | Enrollment to year 1
  Seroconversion in year 1 is defined as a fourfold rise in antibody titers against pathogens of tick-borne disease when comparing titers between baseline and after year 1.
Pathogen seroconversion in study year 2 | Study year 1 to study year 2
  Seroconversion in year 2 is defined as a fourfold rise in antibody titers against pathogens of tick-borne disease when comparing titers between baseline and after year 2.

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Meshnick, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of Rhode Island, Kingston, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A prior study, Tick-borne Illness and Clothing Study (TICS), was conducted in North Carolina by UNC. The current study uses similar methodology as described in the NC study, as it applies to outdoor workers and ticks in the Rhode Island area. — https://clinicaltrials.gov/ct2/show/NCT01454414